CLINICAL TRIAL: NCT01506349
Title: An Assessment of Neurocognitive Symptoms After Gluten Exposure in Adult Patients With Celiac Disease - a Pilot Study
Brief Title: Assessing Neurocognitive Effects of Gluten Exposure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Leffler, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011P000354
Record Dates: First submitted 2011-10-25; First posted 2012-01-10 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Celiac Disease; Neurobehavioral Manifestations
Keywords: celiac disease; gluten; fog; attention
MeSH Terms: conditions — Celiac Disease; Neurobehavioral Manifestations | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crossover Group 1 (Experimental): Group 1 will consume 4 grams of gluten before neurocognitive testing at Visit 2.
  Group 1 will consume placebo before neurocognitive testing at Visit 3.
  Interventions: Dietary Supplement: gluten; Dietary Supplement: Placebo
- Crossover Group 2 (Experimental): Group 2 will consume placebo before neurocognitive testing at Visit 2.
  Group 2 will consume 4 grams of gluten before neurocognitive testing at Visit 3.
  Interventions: Dietary Supplement: gluten; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: gluten — 4 grams of gluten.
Dietary Supplement: Placebo

SUMMARY:
Many patients with celiac disease complain of neurocognitive symptoms such as mental confusion, grogginess, difficulty with concentration and forgetfulness after exposure to gluten. However, there is little data on any possible association between impaired cognitive function and gluten intake in celiac disease. The investigators predict that patients with celiac disease, when exposed to gluten, will experience neurocognitive symptoms such as confusion, forgetfulness and difficulty concentrating.

The goals of this study are to determine the prevalence of neurocognitive symptoms after exposure to gluten in patients with celiac disease and to characterize the nature of these symptoms both in terms of their duration and severity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 18-50 years of age
3. Celiac Disease Group: Positive small intestinal biopsies meeting Marsh II or III histologic criteria for celiac disease at least six months since the time of study entrance as well as positive IgA anti-tissue transglutaminase antibody or positive IgA/IgG anti-Deamidated Gliadin Peptide (DGP) with normal serum IgA
4. Non-Celiac Gluten Sensitive Group: Negative small intestinal biopsies and negative IgA anti-tissue transglutaminase (tTG) or negative IgA/IgG anti-Deamidated Gliadin Peptide (DGP) with normal serum IgA, but with symptomatic response to gluten withdrawal
5. Subject should have well controlled celiac disease and have been on a gluten-free diet for at least six months prior to study enrollment
6. Subject must provide informed consent, as approved by the Institutional Review Board, and agree to complete required study visits, blood work neuropsychological testing and a urine pregnancy test (if applicable).
7. Subject agrees to use appropriate birth control for the duration of the study.

Exclusion Criteria:

1. Subject has other food intolerances or food allergies (other than gluten) that would interfere with the conduct of the study (e.g. corn starch, soy).
2. Subject has a history of severe, acute symptomatic reactions to sporadic gluten ingestion
3. Subject has any chronic active gastrointestinal disease other than celiac disease (e.g. Crohn's disease, irritable bowel syndrome, autoimmune enteropathy, eosinophilic enteritis).
4. Subject should not have daily symptoms concerning for brain fog such as mental confusion or difficulty concentrating, at baseline.
5. Subject has symptomatic neurological or psychiatric disease(s) that would interfere with the conduct of the study.
6. Subject should not have been on corticosteroids or other immunosuppressive agents in the past 3 months.
7. Significant other co-morbidity as determined by the Principal Investigator
8. Subject is deemed inappropriate by the Principal Investigator.
9. Subject is pregnant or breast-feeding at time of participation.
10. Subject weighs less than 110 pounds.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
change in neurocognitive measurements | Baseline, Visit 2 (2 to 6 weeks after baseline), Visit 3 (2 to 6 weeks after Visit 2)
  Neurocognitive measurements will be made using the CogState Research computerized tests

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Leffler, MD, MS, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States